CLINICAL TRIAL: NCT01761097
Title: A Pilot Study to Assess the Role for Endocuff© Assisted Colonoscopy in the Detection of Colonic Cancer and Polyps
Brief Title: Endocuff Adenoma Detection Rate Pilot Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Rob Mead, Dr. R.J.Mead, Cambridge University Hospitals NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: AO92673
Record Dates: First submitted 2013-01-03; First posted 2013-01-04 (Estimated); Last update posted 2013-01-08 (Estimated); Status verified 2013-01

CONDITIONS: Colorectal Adenoma; Colorectal Cancer
Keywords: Adenoma, polyp, colonoscopy.
MeSH Terms: conditions — Colorectal Neoplasms; Adenoma; Polyps

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Endocuff assisted colonoscopy (Active Comparator): Endocuff attachment
  Interventions: Device: Endocuff attachment
- Control standard colonoscopy (Placebo Comparator): Standard colonoscopy

INTERVENTIONS:
Device: Endocuff attachment — Endocuff
  Other Names: ARC endocuff
  Arms: Endocuff assisted colonoscopy

SUMMARY:
Colorectal cancer is the second leading cause of cancer deaths in the UK(1) . Detection of cancer at an early stage, as well as detection and removal of polyps through gold standard colonoscopy examination decreases mortality from the disease. However colonoscopy has a well documented miss rate, with some areas of the bowel difficult to visualise and neoplastic lesions potentially hidden behind folds in the colon.

The Endocuff© is a disposable polymer sleeve with hinged lateral arms. The arms flatten mucosal folds and fix the colonoscope centrally in the bowel lumen allowing controlled withdrawal and improving mucosal visualization. The cap easily attaches to the tip of current colonoscopes without modification. In this single centre, randomised controlled trial, the investigators aim to assess the performance of the current gold standard colonoscopic examination against the current gold standard colonoscopic examination with the Endocuff© attached to the colonoscope.

The investigators aim to recruit 300 patients (150 in each group) who have previously been identified to have colonic polyps or cancers undergoing surveillance colonoscopy following NICE guidelines(2). Colonoscopy will be performed by Joint Advisory Group on gastro-intestinal endoscopy (JAG) certified colonoscopists following quality indicator guidance. All patients undertaking follow up surveillance colonoscopy for previous polyps or cancer will be invited to participate and those agreeing will be randomly allocated to one or other technique.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing surveillance colonoscopy test as part of the colonic adenoma and cancer surveillance programme.
* Ability to understand the nature and requirements of the study and to provide written informed consent.

Exclusion Criteria:

* Contraindication to undergo standard colonoscopy.
* Severe active colitis.
* Known colonic stricture

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2013-01; Primary Completion 2013-10 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with adenomas and cancers detected | immediate

SECONDARY OUTCOMES:
Caecal intubation time | Immediate

OTHER OUTCOMES:
Caecal intubation rate | immediate
Polyp detection rate | immediate

CONTACTS AND LOCATIONS:
Overall Officials: Ewen Cameron, MBBS, Principal Investigator — Cambridge University Hospitals NHS Foundation Trust
Locations (1):
- Addenbrooke's Hospital, Cambridge, United Kingdom